CLINICAL TRIAL: NCT05411913
Title: Immediate Effect of Topical CBD for Musculoskeletal Pain
Brief Title: Topical CBD for Musculoskeletal Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Apothyx, Co. (Industry)
Responsible Party: Principal Investigator, Daniel Charles McShan, PhD, Chief Scientist, Apothyx, Co.
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Topical-CBD-PAIN-001
Record Dates: First submitted 2022-06-02; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — methyl salicylate; Menthol

STUDY DESIGN:
Intervention Model Description: Individuals are provided with a sample of topical substance to apply to a localized region of pain.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Everything is masked by QR code - participant and intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: GoodFOR Pain — GoodFOR Pain is a FDA registered topical analgesic.
Drug: Icy Hot — a FDA OTC registered topical analgesic.
Drug: Tiger Balm — a FDA OTC registered topical analgesic
Drug: Bengay — a FDA OTC registered topical analgesic.
Drug: CBD Clinic Muscle and Joint Pain Relief Ointment — a non FDA registered topical analgesic.
Drug: CBD FX CBD Muscle and Joint Cream: Cooling Formula — a non FDA registered topical analgesic.
Drug: Essential Wholesale Muscle Gel — a non FDA registered topical analgesic.
Drug: Extract Labs Muscle Cream — a non FDA registered topical analgesic.

SUMMARY:
Various OTC and CBD containing topicals are evaluated in a double blind survey. Each sample has a QR code that is to be scanned before applying. The QR code links to a survey form with application instructions and collects participant information and feedback.

ELIGIBILITY:
Inclusion Criteria:

* has Pain

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
Pain Before/After Application | 5 min post intervention
  McGill Pain Questionnaire

SECONDARY OUTCOMES:
Efficiency | 5 min post intervention
  Time and Duration of Pain Relief

IPD SHARING:
Plan to Share IPD: No